CLINICAL TRIAL: NCT00856349
Title: Medtronic Shock-Less Study on Physician Utilization of Shock Reduction Programming
Status: Completed | Type: Observational
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Other Study IDs: Shock-Less
Record Dates: First submitted 2009-02-26; First posted 2009-03-05 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-03 (Estimated); Status verified 2014-07

CONDITIONS: Cardiovascular Disease
Keywords: Implantable Cardioverter Defibrillator (ICD); Cardiac Resynchronization Therapy-Defibrillator (CRT-D); Lead Integrity Alert (LIA); Therapy Programming Report (TPR)
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Analysis cohort: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints.
  Interventions: Behavioral: Therapy Programming Report (TPR)

INTERVENTIONS:
Behavioral: Therapy Programming Report (TPR) — Center-specific therapy programming reports (TPRs) illustrating physician usage of shock reduction programming are provided to each center approximately 9-12 months after their first enrollment and monthly thereafter throughout the study.

SUMMARY:
The purpose of this clinical trial is to determine whether periodic therapy programming reports illustrating physician usage of shock reduction programming can increase utilization of recommended programming guidelines for defibrillators.

DETAILED DESCRIPTION:
Shocks delivered to patients by defibrillators, while life-saving, can create anxiety, pain and decrease quality of life. Previous studies have shown that device programming and features can safely reduce the number of shocks patients receive. This study will explore the extent to which physicians use these programming and features. It will determine whether repeat and frequent awareness to how they program their own subjects and the programming trends of all enrolled subjects will change their programming patterns. This will be accomplished by understanding physicians' device programming behaviors and providing reports as a tool to help physicians manage their subjects and provide shock reduction programming recommended by previous publications.

ELIGIBILITY:
Inclusion Criteria:

* Subject (or subject's legally authorized representative) is willing and able to sign and date the Patient Consent Form (PCF) and authorization for access to and use of health information, if applicable
* Subject has been implanted with a Medtronic market released ICD or CRT-D device (US/Canada - Concerto®/Virtuoso® or newer model; AsiaPacific, Israel, Latin America - EnTrust™, InSync Sentry®, or Concerto®/Virtuoso® or newer model) within the past 30 days
* Subject has commercially released RA (if applicable), RV, and LV (if applicable) leads

Exclusion Criteria:

* Subject is enrolled in a concurrent study that has not been approved for concurrent enrollment by the Medtronic Clinical Trial Leader

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects implanted with a Medtronic market released single, dual, or triple chamber defibrillator (US/Canada - Concerto®/Virtuoso® or newer model; AsiaPacific, Israel, Latin America - EnTrust™, InSync Sentry®, or Concerto®/Virtuoso® or newer model) within the past 30 days are eligible for participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 4384 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Silver, M.D., Principal Investigator — Raleigh Cardiology Associates
Locations (104):
- United States (83):
  - Anniston, Alabama
  - Phoenix, Arizona
  - Tucson, Arizona
  - Hot Springs, Arkansas
  - Little Rock, Arkansas
  - Fremont, California
  - Fresno, California
  - Modesto, California
  - Northridge, California
  - Orange, California
  - San Bernardino/Los Angeles, California
  - Ventura, California
  - New Haven, Connecticut
  - Fort Lauderdale, Florida
  - Jacksonville, Florida
  - Ocala, Florida
  - Palm Beach Gardens, Florida
  - Pensacola, Florida
  - Plantation, Florida
  - Rockledge, Florida
  - St. Petersburg, Florida
  - Zephyrhills, Florida
  - Atlanta, Georgia
  - Berwyn, Illinois
  - Elk Grove Village, Illinois
  - Maywood, Illinois
  - Evansville, Indiana
  - Fort Wayne, Indiana
  - Scarborough, Maine
  - Baltimore, Maryland
  - Takoma Park, Maryland
  - New Bedford, Massachusetts
  - Flint, Michigan
  - Kalamazoo, Michigan
  - Lansing, Michigan
  - Saint Joseph, Michigan
  - Robbinsdale, Minnesota
  - Saint Louis Park, Minnesota
  - Jackson, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Las Vegas, Nevada
  - Cherry Hill, New Jersey
  - Clifton, New Jersey
  - Flemington, New Jersey
  - Newark, New Jersey
  - Albuquerque, New Mexico
  - Elmira, New York
  - Flushing, New York
  - New York, New York
  - Utica, New York
  - Williamsville, New York
  - Charlotte, North Carolina
  - Raleigh, North Carolina
  - Wilmington, North Carolina
  - Winston-Salem, North Carolina
  - Fargo, North Dakota
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Mansfield, Ohio
  - Youngstown, Ohio
  - Lawton, Oklahoma
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Erie, Pennsylvania
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Sioux Falls, South Dakota
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - El Paso, Texas
  - Fort Sam Houston, Texas
  - Houston, Texas
  - McAllen, Texas
  - Tyler, Texas
  - Charlottesville, Virginia
  - Manassas, Virginia
  - Charleston, West Virginia
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Buenos Aires, Argentina
- Australia (3):
  - Adelaide, South Australia
  - Frankston, Victoria
  - Perth, Western Australia
- Canada (7):
  - Edmonton, Alberta
  - Victoria, British Columbia
  - Winnipeg, Manitoba
  - Kitchener, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Sherbrooke, Quebec
- China (2):
  - Guangzhou, Guangdong
  - Beijing
- Kowloon, Hong Kong
- India (2):
  - New Dehli, National Capital Territory of Delhi
  - Saket, New Dehli
- Mexico City, Mexico
- Frankton, Hamilton, New Zealand
- Singapore, Singapore
- Seoul, South Korea
- Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Joung B, Lexcen DR, Ching CK, Silver MT, Piccini JP, Sterns LD, Rabinovich R, Pickett RA, Liu S, Brown ML, Cheng A. Additional antitachycardia pacing programming strategies further reduce unnecessary implantable cardioverter-defibrillator shocks. Heart Rhythm. 2020 Jan;17(1):98-105. doi: 10.1016/j.hrthm.2019.07.027. Epub 2019 Jul 29. PMID 31369873

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the Shock-Less study between April 2009 and January 2012 from 118 centers worldwide in North America, Central/South America, Australia/New Zealand and Asia.
Pre-assignment Details: A total of 252 (6%) out of the 4384 enrolled subjects were excluded from the analysis cohort due to the following reasons: baseline device interrogation not available (217/252; 86%), inclusion/exclusion criteria not met (16/252, 6%), indication for ICD implant not specified (11/252; 4%), and VF therapy/detection not turned ON (8/252; 3%).
Groups:
- Analysis Cohort: Enrolled subjects who met study eligibility criteria and contributed data toward the primary and/or secondary study endpoints.
Period: Overall Study
Arm/Group | Analysis Cohort
Started | 4132
12 Month Follow-up | 3228
18 Month Follow-up | 2467
24 Month Follow-up | 1698
Completed | 3111
Not Completed | 1021
Not completed — Death | 418
Not completed — Withdrawal by Subject | 116
Not completed — Lost to Follow-up | 91
Not completed — Protocol Violation | 38
Not completed — Physician Decision | 13
Not completed — Subject relocation | 104
Not completed — Device explant | 33
Not completed — Site closure | 78
Not completed — Subject changed Dr, insurance issue, etc | 130

BASELINE CHARACTERISTICS:
Population: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints.
Arm/Group | Analysis Cohort
Number analyzed (Participants) | 4132
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 971
  Male | 3161
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 14
  Asian | 295
  Native Hawaiian or Other Pacific Islander | 9
  Black or African American | 360
  White | 3151
  More than one race | 5
  Unknown or Not Reported | 298
Region of Enrollment [Number; unit: participants]
  United States | 3307
  Taiwan | 27
  Hong Kong | 15
  Mexico | 8
  Canada | 434
  Argentina | 19
  Singapore | 39
  Australia | 69
  New Zealand | 26
  China | 28
  Korea, Republic of | 24
  India | 118
  Thailand | 18

OUTCOME MEASURES:

1. Primary Outcome: Change in Shock Reduction Programming Adoption
Description: Change in percentage of subjects programmed to evidence-based target from baseline (pre-TPR distribution) to last follow-up (post-TPR distribution).
  Shock-reduction programming parameters:
  LIA (Lead Integrity Alert): Uploadable algorithm with the ability to increase the time between a lead fracture and potential delivery of an unnecessary shock.
  SVT (Supraventricular Tachycardia) Limit: The maximum cycle length that Wavelet and PR logic will be applied to arrhythmias.
  VF NID PP: Number of intervals to detect (NID) an arrhythmia in the VF zone for primary prevention (PP) patients.
  VF NID SP: Number of intervals to detect (NID) an arrhythmia in the VF zone for secondary prevention (SP) patients.
  Wavelet: Discriminator to help determine if arrhythmia is ventricular or supraventricular in single chamber ICDs.
  PR Logic: Discriminator to help determine if arrhythmia is ventricular or supraventricular in dual chamber ICDs and CRT-Ds.
Time Frame: Overall study (20 months on average)
Population: Subjects with paired baseline and follow-up programming data
Measure: Number; unit: percentage of participants
Groups:
- Subjects With Paired Programming Data: Subjects with paired baseline and follow-up programming data to evaluate changes in shock-reduction programming parameters
Arm/Group | Subjects With Paired Programming Data
Number analyzed (Participants) | 2201
percentage of participants
  Increase in % on target (LIA) | 13.6
  Increase in % on target (SVT Limit) | 6.8
  Increase in % on target (VF NID PP) | 9.0
  Increase in % on target (VF NID SP) | 3.5
  Increase in % on target (Wavelet) | 9.5
  Increase in % on target (PR Logic) | 3.2
Statistical Analysis 1: Comparison: Subjects With Paired Programming Data; LIA (Lead Integrity Alert): Uploadable algorithm with the ability to increase the time between a lead fracture and potential delivery of an unnecessary shock; Test type: Superiority or Other; p < 0.0001, McNemar; Increase in % on target (LIA) = 13.6
Statistical Analysis 2: Comparison: Subjects With Paired Programming Data; SVT (Supraventricular Tachycardia) Limit: The maximum cycle length that Wavelet and PR logic will be applied to arrhythmias; Test type: Superiority or Other; p < 0.0001, McNemar; Increase in % on target (SVT Limit) = 6.8
Statistical Analysis 3: Comparison: Subjects With Paired Programming Data; VF NID PP: Number of intervals to detect (NID) an arrhythmia in the VF zone for primary prevention (PP) patients; Test type: Superiority or Other; p < 0.0001, McNemar; Increase in % on target (VF NID PP) = 9.0
Statistical Analysis 4: Comparison: Subjects With Paired Programming Data; VF NID SP: Number of intervals to detect (NID) an arrhythmia in the VF zone for secondary prevention (SP) patients; Test type: Superiority or Other; p = 0.0116, McNemar; Increase in % on target (VF NID SP) = 3.5
Statistical Analysis 5: Comparison: Subjects With Paired Programming Data; Wavelet: Discriminator to help determine if arrhythmia is ventricular or supraventricular in single chamber ICDs; Test type: Superiority or Other; p < 0.0001, McNemar; Increase in % on target (Wavelet) = 9.5
Statistical Analysis 6: Comparison: Subjects With Paired Programming Data; PR Logic: Discriminator to help determine if arrhythmia is ventricular or supraventricular in dual chamber ICDs and CRT-Ds; Test type: Superiority or Other; p < 0.0001, McNemar; Increase in % on target (PR Logic) = 3.2

2. Secondary Outcome: Lead Integrity Alert (LIA) Performance
Description: Causes for LIA triggers reported during the study
Time Frame: Overall study (20 months on average)
Population: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints.
Measure: Number; unit: percentage of subjects with LIA triggers
Units Other Than Participants: Subjects who experienced LIA triggers
Arm/Group | Analysis Cohort
Number analyzed (Participants) | 4132
Number analyzed (Subjects who experienced LIA triggers) | 23
percentage of subjects with LIA triggers
  Lead fracture | 30.4
  Dislodgment | 8.7
  Connector issure | 8.7
  RV lead noise | 8.7
  VT/VF | 8.7
  EMI | 4.3
  Oversensing undefined | 17.4
  Unknown | 17.4

3. Secondary Outcome: Reasons for Inappropriate Shocks
Description: Reasons for inappropriate shocks observed during the study
Time Frame: Overall study (20 months on average)
Population: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints.
Measure: Number; unit: percentage of inappropriate shocks
Units Other Than Participants: inappropriate shocks
Arm/Group | Analysis Cohort
Number analyzed (Participants) | 4132
Number analyzed (inappropriate shocks) | 553
percentage of inappropriate shocks
  AF/AFL | 56.4
  Other SVT (sinus tach, atrial tach, etc.) | 29.5
  T-wave oversensing | 6.9
  Oversensing due to lead noise | 6.0
  Non-Sustained VT | 0.5
  Other | 0.7

4. Secondary Outcome: Actions Taken Following a Shock
Description: Characterization of actions taken by the subject immediately following a device shock
Time Frame: Overall study (20 months on average)
Population: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints.
Measure: Number; unit: percentage of subjects with shocks
Units Other Than Participants: Subjects who experienced shocks
Arm/Group | Analysis Cohort
Number analyzed (Participants) | 4132
Number analyzed (Subjects who experienced shocks) | 421
percentage of subjects with shocks
  ER visit | 28
  Called follow-up clinic | 23
  Clinic visit | 12.4
  CareLink transmission | 6.7
  Off-hours follow-up clinician call | 2.6
  Urgent Care visit | 0.7
  Other | 10.2
  No action taken | 29

5. Secondary Outcome: Barriers to Utilization of Shock Reduction Programming
Description: Characterization of barriers to physician utilization of shock reduction programming
Time Frame: 24 months follow-up visit
Population: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints.
Measure: Number; unit: % of subjects not programmed to target
Units Other Than Participants: Subjects not programmed to target
Arm/Group | Analysis Cohort
Number analyzed (Participants) | 1698
Number analyzed (Subjects not programmed to target) | 27
% of subjects not programmed to target
  Physician preference | 51.9
  Medical history | 7.4
  Current subject condition | 3.7
  Utilization of nominal settings | 3.7
  Not reported | 37

6. Secondary Outcome: Relationship of Subject Characteristics and Geographical Regions With Shock Reduction Programming Utilization
Description: Characterization of shock reduction programming utilization by subject characteristics and geographical regions
Time Frame: Overall study (20 months on average)
Population: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints, with final programming data available post-TPR distribution.
Measure: Number; unit: percentage of participants
Groups:
- Subjects With Final Programming Data Available: Enrolled subjects who met study eligibility criteria and contributed data toward study endpoints, with final programming data available post-TPR distribution.
Arm/Group | Subjects With Final Programming Data Available
Number analyzed (Participants) | 3714
percentage of participants
  VF NID PP % on target - Male | 31.6
  VF NID PP % on target - Female | 30.2
  VF NID PP % on target - North America | 31.1
  VF NID PP % on target - Asia | 31.2
  VF NID PP % on target - ANZ | 40.3
  VF NID PP % on target - Central/South America | 11.1

ADVERSE EVENTS:
Description: Adverse events were not collected in this study
Arm/Group | Analysis Cohort
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, contracts allow investigators to publish study results per the protocol and publication plan. Investigators and Participating Institutions will provide any publication of Study Data generated by PI and/or Participating Institution to Medtronic for review prior to submission to determine if confidential information ("CI") is included and to check for technical correctness. Medtronic may not censor/interfere with the publication beyond the extent necessary to protect CI.